CLINICAL TRIAL: NCT00856583
Title: Sertindole Versus Risperidone Safety Outcome Study: a Randomised, Partially-blinded, Parallel-group, Active-controlled, Post-marketing Study
Brief Title: Safety Study of Sertindole Versus Risperidone Under Normal Conditions of Use
Acronym: SCoP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 99824; 2004-000213-19 (EudraCT Number)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2011-08-01 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertindole (Experimental): Normally in the range of 4 to 20 mg/day
  Interventions: Drug: Sertindole
- Risperidone (Active Comparator): Normally in the range of 2 to 8 mg/day
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Sertindole — Sertindole was supplied as 4, 12, 16, and 20 mg tablets. The start and maintenance dosages as well as dose titration were set by the investigator, in accordance with the national Summary of Product Characteristics (SPC) for sertindole; in countries where sertindole was not marketed, the European Union (EU) SPC applied (all national and EU SPCs were essentially identical). Recommended dose range: 12 to 20 mg/day. The investigators were instructed to contact H. Lundbeck A/S if they deemed it necessary to increase the dose of sertindole to 24 mg/day, which was allowed in exceptional cases
  Other Names: Serdolect
  Arms: Sertindole
Drug: Risperidone — Risperidone was supplied as 1, 2, 3, and 4 mg tablets. The start and maintenance dosages as well as dose titration were set by the investigator, in accordance with the national SPC for risperidone. Recommended dose range: 2 to 8 mg/day
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
The purpose of the study is to determine whether there is an increased all-cause mortality in sertindole-treated patients in comparison to patients treated with a well-known antipsychotic (risperidone) when used under normal marketed conditions in the treatment of schizophrenia.

DETAILED DESCRIPTION:
The Committee for Medicinal Products for Human Use (CHMP) requested a post-marketing study to ascertain that the favourable benefit-risk profile and low mortality rates seen in the clinical studies with sertindole would not be offset by higher mortality rates when sertindole was used under more normal conditions of use. It was recognised that, in a clinical trial setting, strict patient selection and monitoring could lead to higher compliance in patient management and thereby to a lower mortality rate. Study 99824 was therefore designed in collaboration with the CHMP as an open-label, randomised study with minimum study management that focused on mortality and general patient safety. The duration of the treatment period was not fixed. No efficacy measures were included.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed the Informed Consent Form or, if he/she is not able to sign it (according to the ICH GCP guidelines and the Declaration of Helsinki), the patient's legal representative has signed the Informed Consent Form
* The patient has been diagnosed with schizophrenia
* Based on the patient's clinical status, new or change of antipsychotic treatment is indicated
* The patient is at least 18 years of age
* The patient meets the criteria set out in the national SPCs for sertindole and risperidone. For those countries in which sertindole was not marketed, the EU SPC applied

Exclusion Criteria:

* The last treatment taken by the patient was sertindole or risperidone
* The patient has never previously received any antipsychotic drug therapy
* The patient has contraindications to treatment with either sertindole or risperidone
* In addition to sertindole/risperidone, treatment with another antipsychotic is indicated
* The patient is homeless
* The patient has previously been included in one of the two H. Lundbeck A/S post-marketing studies, 99823 or 99824
* The patient is, in the opinion of the investigator, unlikely to comply with the study protocol or unsuitable for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9809 (Actual)
Dates: Start 2002-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Peuskens J, Tanghoj P, Mittoux A; Sertindole Cohort. The Sertindole Cohort Prospective (SCoP) study: rationale, design and methodology. Pharmacoepidemiol Drug Saf. 2008 May;17(5):425-33. doi: 10.1002/pds.1594. PMID 18384186
- [Result] Thomas SH, Drici MD, Hall GC, Crocq MA, Everitt B, Lader MH, Le Jeunne C, Naber D, Priori S, Sturkenboom M, Thibaut F, Peuskens J, Mittoux A, Tanghoj P, Toumi M, Moore ND, Mann RD. Safety of sertindole versus risperidone in schizophrenia: principal results of the sertindole cohort prospective study (SCoP). Acta Psychiatr Scand. 2010 Nov;122(5):345-55. doi: 10.1111/j.1600-0447.2010.01563.x. PMID 20384598
- [Result] Crocq MA, Naber D, Lader MH, Thibaut F, Drici M, Everitt B, Hall GC, Le Jeunne C, Mittoux A, Peuskens J, Priori S, Sturkenboom M, Thomas SH, Tanghoj P, Toumi M, Mann R, Moore ND. Suicide attempts in a prospective cohort of patients with schizophrenia treated with sertindole or risperidone. Eur Neuropsychopharmacol. 2010 Dec;20(12):829-38. doi: 10.1016/j.euroneuro.2010.09.001. PMID 20926264
- [Result] De Hert M, Mittoux A, He Y, Peuskens J. Metabolic parameters in the short- and long-term treatment of schizophrenia with sertindole or risperidone. Eur Arch Psychiatry Clin Neurosci. 2011 Jun;261(4):231-9. doi: 10.1007/s00406-010-0142-x. Epub 2010 Sep 5. PMID 20820795
- [Result] De Hert M, Mittoux A, He Y, Peuskens J. A head-to-head comparison of sertindole and risperidone on metabolic parameters. Schizophr Res. 2010 Nov;123(2-3):276-7. doi: 10.1016/j.schres.2010.07.030. Epub 2010 Aug 21. No abstract available. PMID 20732794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 593 centres in 38 countries (Europe and Asia). First patient first visit: 11 July 2002. Last patient last visit: 22 February 2008.
Period: Overall Study
Arm/Group | Sertindole | Risperidone
Started | 4905 (Patients treated) | 4904 (Patients treated)
Completed | 1768 (Patients who were still on study drug at the time of study closure) | 2307 (Patients who were still on study drug at the time of study closure)
Not Completed | 3137 | 2597
Not completed — Lack of Efficacy | 389 | 377
Not completed — Serious Adverse Event (SAE) | 99 | 65
Not completed — Non-SAE: Mostly Asymptomatic ECGs | 393 | 179
Not completed — Non-compliance | 305 | 262
Not completed — Withdrawal by Subject | 1092 | 919
Not completed — Physician Decision | 59 | 82
Not completed — Pregnancy | 14 | 5
Not completed — Other | 92 | 104
Not completed — Non-evaluable: Patient on Polytherapy | 694 | 604

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertindole | Risperidone | Total
Number analyzed (Participants) | 4905 | 4904 | 9809
Age Continuous [Mean (Standard Deviation); unit: years] | 38.4 (11.8) | 38.3 (11.7) | 38.3 (11.8)
Age, Customized [Number; unit: participants]
  18 to 65 years | 4806 | 4820 | 9626
  > 65 years | 99 | 84 | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2195 | 2188 | 4383
  Male | 2710 | 2716 | 5426
Duration of schizophrenia [Number; unit: participants]
  Unknown | 125 | 87 | 212
  < 5 years | 1450 | 1468 | 2918
  5 to 10 years | 1254 | 1278 | 2532
  > 10 years | 2076 | 2071 | 4147
Reasons for prescription of study drug [Number; unit: participants]
  Adverse drug reaction | 1121 | 1072 | 2193
  Lack of efficacy | 2542 | 2580 | 5122
  None or poor compliance | 161 | 169 | 330
  Patient's choice | 992 | 979 | 1971
  Other | 89 | 104 | 193
Number of previous suicide attempts [Number; unit: participants]
  Unknown | 17 | 11 | 28
  0 previous suicide attempts | 4281 | 4288 | 8569
  1 previous suicide attempt | 378 | 377 | 755
  2 previous suicide attempts | 125 | 126 | 251
  3 previous suicide attempts | 52 | 53 | 105
  4 previous suicide attempts | 18 | 13 | 31
  >= 5 previous suicide attempts | 34 | 36 | 70
Time since last suicide attempt [Number; unit: participants]
  No previous suicide attempt or unknown | 4298 | 4301 | 8599
  < 1 year | 122 | 117 | 239
  1 to 5 years | 226 | 218 | 444
  > 5 years | 259 | 268 | 527

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Mortality
Description: The analysis was based on all deaths from the Whole Randomised Treatment (WRT)+30 days period and the Only Randomised Treatment (ORT) period, respectively
Time Frame: As study design allowed patients to continue study drug until the study was closed, many patients were followed for several years, with an overall median time period of approximately 14 months
Population: The analysis population included all patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants
  Number of deaths (WRT+30 days) | 64 | 61
  Number of deaths (ORT) | 40 | 44
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; The basis for the statistical analysis of the first primary outcome was the null hypothesis of an excess mortality in sertindole-treated patients compared to the mortality in risperidone-treated patients for the WRT+30 days period; Test type: Non-Inferiority or Equivalence — If the upper limit of the 90% confidence interval (CI) for the estimated all-cause mortality ratio was <1.5 (pre-specified), the null hypothesis was rejected. With this limit, 7,600 patient years of exposure (PYE) were required to ensure 80% power at the 5% significance level of rejecting the null hypothesis when assuming a mortality of 2 deaths per 100 PYE. As the actual mortality was only about half that anticipated, more exposure was necessary and the duration of the study increased markedly; p = 0.05, Cox Proportional Hazard; Adjusted for: age, sex, time since last suicide attempt, last previous antipsychotic treatment (mono-/polytherapy), year since start of enrollment; Hazard Ratio (HR) = 1.117, 90% CI 2-sided [0.831 to 1.500] — The hazard ratio is calculated as sertindole (numerator) versus risperidone (denominator)
Statistical Analysis 2: Comparison: Sertindole vs Risperidone; The basis for the statistical analysis of the first primary outcome was the null hypothesis of an excess mortality in sertindole-treated patients compared to the mortality in risperidone-treated patients for the ORT period; Test type: Non-Inferiority or Equivalence — If the upper limit of the 90% CI for the estimated all-cause mortality ratio was <1.5 (pre-specified), the null hypothesis was rejected. With this limit, 7,600 PYE were required to ensure 80% power at the 5% significance level of rejecting the null hypothesis when assuming a mortality of 2 deaths per 100 PYE. As the actual mortality was only about half that anticipated, more exposure was necessary and the duration of the study increased markedly; p < 0.05, Cox Proportional Hazard; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.980, 90% CI 2-sided [0.684 to 1.405] — The hazard ratio is calculated as sertindole (numerator) versus risperidone (denominator)

2. Secondary Outcome: Cause-specific Mortality: Number of Participants With Cardiac Deaths - ISC
Description: The analysis was based on all deaths from the WRT+30 days period using the classification performed by the ISC.
  The ISC reviewed and classified those adverse events which resulted in death or hospitalisation or were possible suicide attempts and this review was blinded to exposure. The definition of cardiac death was intentionally wide; sudden or unexplained deaths were assumed to be cardiac if there was no non-cardiac explanation. To ensure consistent evaluation and classification, the ISC decided a priori to classify all instances of self harm as possible suicide.
Time Frame: as for outcome 1
Population: The analysis population included all patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 31 | 12
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; The basis for the statistical analysis of this secondary outcome was the null hypothesis of mortality hazard ratio equal to 1 for the sertindole-treated patients versus risperidone-treated patients during the WRT+30 days period; Test type: Superiority or Other; p = 0.0022, Cox Proportional Hazard; Adjusted: age, sex, time since last suicide attempt, last previous antipsychotic treatment (mono-/polytherapy), region, year since start of enrollment; Hazard Ratio (HR) = 2.84, 95% CI 2-sided [1.45 to 5.55]

3. Primary Outcome: Second Primary Outcome: Number of Participants With Cardiac Events, Including Arrhythmias, Requiring Hospitalisation
Description: Second primary endpoint: a serious adverse event where the patient was hospitalised and for which the Independent Safety Committee (ISC) classified the event as a cardiac event with documented arrhythmia. The analysis of this outcome was not performed due to low number of events. The presented analysis is a replacement analysis using all cardiac events, including arrhythmias, that required hospitalisation
Time Frame: as for outcome 1
Population: The analysis population included all patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 10 | 6
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; The basis for the statistical analysis of time to 1st occurence of the secondary primary outcome (one patient in the risperidone group reported more than one occurrence of this event) was the null hypothesis of hazard ratio equal to 1 for the sertindole-treated patients versus risperidone-treated patients during the WRT+30 days period; Test type: Superiority or Other; p = 0.29, Cox Proportional Hazard; Adjusted for: age and sex; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [0.63 to 4.78]

4. Secondary Outcome: Cause-specific Mortality: Number of Participants With Completed Suicides - ISC
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 14 | 21
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.34, Cox Proportional Hazard; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.36 to 1.41]

5. Secondary Outcome: Cause-specific Mortality: Number of Participants With Other Than Cardiac Deaths and Completed Suicides - ISC
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 19 | 28
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.26, Cox Proportional Hazard; Adjusted for: age, sex, last previous antipsychotic treatment (mono-/polytherapy), year since start of enrollment; Hazard Ratio (HR) = 0.715, 95% CI 2-sided [0.40 to 1.28]

6. Secondary Outcome: Cause-specific Mortality: Number of Participants With Cardiac Deaths - MedDRA
Description: The analysis was based on all deaths from the WRT+30 days period using the classification based upon the Medical Dictionary for Regulatory Activities (MedDRA) terminology, that is, as reported by the investigator
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 17 | 8
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.081, Cox Proportional Hazard; Adjusted for: age, sex, last previous antipsychotic treatment (mono-/polytherapy); Hazard Ratio (HR) = 2.13, 95% CI 2-sided [0.91 to 4.98]

7. Secondary Outcome: Cause-specific Mortality: Number of Participants With Completed Suicides - MedDRA
Description: The analysis was based on all deaths from the WRT+30 days period using the classification based upon MedDRA terminology, that is, as reported by the investigator
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 13 | 21
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.24, Cox Proportional Hazard; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.33 to 1.32]

8. Secondary Outcome: Cause-specific Mortality: Number of Participants With Other Than Cardiac Deaths and Completed Suicides - MedDRA
Description: as for outcome 7
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 34 | 32
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.59, Cox Proportional Hazard; Adjusted for: age, sex, last previous antipsychotic treatment (mono-/polytherapy), year since start of enrollment; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.70 to 1.85]

9. Secondary Outcome: Number of Participants With Suicide Attempts (Fatal and Non-fatal) - ISC
Description: The analysis was based on all suicides and suicide attempts from the WRT+30 days period using the classification performed by the ISC.
  The ISC reviewed and classified those adverse events which resulted in death or hospitalisation or were possible suicide attempts and this review was blinded to exposure. The definition of cardiac death was intentionally wide; sudden or unexplained deaths were assumed to be cardiac if there was no non-cardiac explanation. To ensure consistent evaluation and classification, the ISC decided a priori to classify all instances of self harm as possible suicide.
Time Frame: as for outcome 1
Population: The analysis population included all patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 68 | 76
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; The basis for the statistical analysis of time to 1st occurence of this secondary outcome was the null hypothesis of hazard ratio equal to 1 for the sertindole-treated patients versus risperidone-treated patients during the WRT+30 days period; Test type: Superiority or Other; p = 0.65, Cox Proportional Hazard; Adjusted for: age, sex, duration of schizophrenia, time since last suicide attempt, year since start of enrollment; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.66 to 1.29]

10. Secondary Outcome: Number of Participants With Suicide Attempts (Fatal and Non-fatal) - MedDRA
Description: The analysis was based on all suicides and suicide attempts from the WRT+30 days period using the classification based upon MedDRA terminology, that is, as reported by the investigator
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 43 | 65
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.044, Cox Proportional Hazard; Adjusted for: age, sex, duration of schizophrenia, time since last suicide attempt, year since start of enrollment; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.45 to 0.99]

11. Secondary Outcome: Number of Participants With Hospitalisations, Excluding Hospitalisations Related to the Primary Psychiatric Disease
Description: The analysis was based on time from start of study drug to first hospitalisation during the WRT+30 days period
Time Frame: as for outcome 1
Population: The analysis population included all patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 174 | 149
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.040, Cox Proportional Hazard; Adjusted for: age, sex, time since last suicide attempt, last antipsychotic medication (a-/typicals/both), region, year since start of enrollment; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [1.01 to 1.57]

12. Secondary Outcome: Number of Participants With Discontinuation of Treatment for Any Reason Other Than Study Closure
Description: The analysis was based on time from start of study drug until stop of study drug for any reason other than sponsor closure of the study
Time Frame: as for outcome 1
Population: The analysis population included all patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sertindole | Risperidone
Number analyzed (Participants) | 4905 | 4904
participants | 3136 (430 PET?) | 2597 (433)
Statistical Analysis 1: Comparison: Sertindole vs Risperidone; The basis for the statistical analysis of this secondary outcome was the null hypothesis of hazard ratio equal to 1 for the sertindole-treated patients versus risperidone-treated patients during the WRT+30 days period; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazard; Adjusted: disease duration, time since last suicide attempt, last antipsychotic medication (a-/typicals/both), region, year since start of enrollment; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.28 to 1.43]

ADVERSE EVENTS:
Time Frame: As study design allowed patients to continue study drug until the study was closed, many patients were followed for several years, with an overall median time period of approximately 14 months.
Description: Data on all serious adverse events and non-serious cardiac adverse events were collected.
Arm/Group | Sertindole | Risperidone
Serious Adverse Events (participants affected / at risk) | 266/4905 | 217/4904
Other Adverse Events (participants affected / at risk) | 397/4905 | 11/4904
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertindole (N=4905) | Risperidone (N=4904)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (2)
Arrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperprolactinaemia (Endocrine disorders) | 3 (3) | 3 (3)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 2 (2)
Eyelid disorder (Eye disorders) | 1 (1) | 0 (0)
Meibomianitis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 12 (12) | 2 (2)
Drowning (General disorders) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sudden death (General disorders) | 1 (1) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular damage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infection in an immunocompromised host (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (9) | 7 (7)
Pneumonia chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 4 (4) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Vaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 21 (23) | 14 (16)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 15 (16) | 8 (8)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Self mutilation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 17 (18) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Medical observation (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetis mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Scrotal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Brain damage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4) | 5 (6)
Diabetic coma (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 5 (5) | 3 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 2 (2) | 2 (2)
Neuroleptic malignant syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 13 (13) | 21 (21)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 3 (3) | 3 (3)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 7 (7) | 4 (4)
Suicide attempt (Psychiatric disorders) | 29 (30) | 45 (49)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Haematosalpinx (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)
Drug abuser (Social circumstances) | 1 (1) | 0 (0)
Physical assault (Social circumstances) | 1 (1) | 1 (1)
Social problem (Social circumstances) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Plastic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sertindole (N=4905) | Risperidone (N=4904)
Electrocardiogram QT prolonged (Investigations) | 397 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the investigator will be subject to mutual agreement between the investigator and H. Lundbeck A/S.